CLINICAL TRIAL: NCT03470103
Title: A Prospective Observational Study in Patients With Wet Age-related Macular Degeneration or Diabetic Macular Edema to Assess the freQuency of Use of Intravitreal Aflibercept in Routine Clinical Practices in Latin America
Brief Title: A Study in Patients With Wet Age-related Macular Degeneration or Diabetic Macular Edema to Assess the freQuency of Use of Intravitreal Aflibercept in Routine Clinical Practices in Latin America
Acronym: AQUILA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19518
Record Dates: First submitted 2018-02-05; First posted 2018-03-19 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Macular Degeneration
Keywords: Wet age-related macular degeneration(wAMD); Diabetic macular edema(DME)
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Treatment naïve wAMD: The decision regarding treatment is made at the discretion of the attending physician, according to his/her medical practice
  Interventions: Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321)
- Treatment naïve DME: The decision regarding treatment is made at the discretion of the attending physician, according to his/her medical practice
  Interventions: Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321)
- Previously treated wAMD: The decision regarding treatment is made at the discretion of the attending physician, according to his/her medical practice
  Interventions: Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321)
- Previously treated DME: The decision regarding treatment is made at the discretion of the attending physician, according to his/her medical practice
  Interventions: Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321) — Use of intravitreal aflibercept in routine clinical practice in Latin America

SUMMARY:
The main objectives of this observational cohort study are to describe the use of intravitreal aflibercept and to describe follow-up as well as treatment patterns in patients with wAMD or DME in routine clinical practice in Latin America for a study population of treatment naive patients and those who have received prior therapy (anti-VEGF injections, laser, steroids, etc.) and are being switched to intravitreal aflibercept injection.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years of age for DME patients,
* Age: ≥55 for wAMD patients
* Decision to treat with intravitreal aflibercept in the study eye prior to patient enrolment as per the physician's routine clinical practice and following the local Product monograph recommendations. Patients who are treatment naïve (no previous intravitreal treatment received, including, anti- VEGF agents, steroids, steroid implants and/or PDT) and patients that are switching from a different anti-VEGF therapy are both eligible to be included. DME patients that have received previous laser only will be classified as treatment naïve.
* If of childbearing potential, female willing to use effective contraception during treatment and for at least 3 months after the last intravitreal injection of aflibercept

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice.
* Patients currently being treated with intravitreal aflibercept in the study eye.
* Patients who are hypersensitive to this drug, to any ingredient in the formulation, or to any component of the container. For a complete listing, see the DOSAGE FORMS, COMPOSITION AND PACKAGING section of the local product monograph.
* Ocular or peri-ocular infection in either eye.
* Active intraocular inflammation in the study eye.
* Scar, fibrosis, or atrophy involving the center of the fovea in the study eye.
* Patients with advanced glaucoma, visually significant cataracts, or any eye disease likely to require surgery during the study period in the study eye.
* Concomitant ocular or systemic administration of drugs that could interfere with or potentiate the mechanism of action of intravitreal aflibercept, including anti-VEGF agents.
* Patients receiving a different anti-VEGF agent other than intravitreal aflibercept for the fellow eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with wAMD or DME treated with intravitreal aflibercept. If both eyes are eligible, data from both eyes will be captured, but only one eye will be considered the study eye and included in the study analyses. The eye included will be at the physician's discretion and only visits related to the study eye will be captured in the electronic Case Report Form (eCRF).
Sampling Method: Non-Probability Sample
Enrollment: 643 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Mean change of visual acuity as measured by ETDRS or Snellen chart | At baseline and 12 months
  ETDRS: Early treatment diabetic retinopathy study

SECONDARY OUTCOMES:
Mean change in visual acuity as measured by ETDRS or Snellen chart | At baseline and 12 months
  Mean change in visual acuity between baseline and 12 months for the overall population (treatment naïve + previously treated patients) by indication, wAMD and DME.
Change in retinal thickness as measured by OCT | At baseline and 12 months
  OCT: Optical coherence tomography
Mean time between injections by indication | Up to 12 months
Mean number of injections by indication | At 12 months
Duration of previous treatments by indication | Up to 12 months
  In the previously treated subpopulation
Type (anti-VEGF, laser, steroids, etc) of previous treatments by indication | Up to 12 months
  In the previously treated subpopulation
Percentage of patients with no fluid determined by OCT | At 12 months
  Absence of fluid includes all types of fluid and would be determined by physicians judgment
Percentage of patients achieving a Snellen equivalent of 20/40 or better | At 12 months
  About 70 ETDRS(Early treatment diabetic retinopathy study) letters
Percentage of patients gaining ≥15 ETDRS letter | At 12 months
Presence/absence of pigment epithelium detachments (PED) | At 12 months
  In the wAMD population
Number of adjunctive therapies | At 12 months
  In the DME population
Type of adjunctive therapies based on medical records or on interviewing the patient | At 12 months
Diabetic retinopathy severity (mild, moderate, severe) | At 12 months
  In the DME population
Reason to switch to intravitreal aflibercept based on medical records or on interviewing the patient | At 12 months
Number of monitoring visits | At 12 months
  Visits only for diagnostic purposes, but without injections
Number of combined visits | At 12 months
  Visits for monitoring and injection
Number of visits outside the study center | At 12 months
  Visits with other non-ophthalmology specialists, i.e. endocrinologists, family physician, etc.
Number of optical coherence tomography (OCT) assessments per patient | At 12 months
Number of visual acuity tests | At 12 months
Number of fundoscopy examinations | At 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- Many locations, Multiple Locations, Argentina
- Many locations, Multiple Locations, Colombia
- Many locations, Multiple Locations, Costa Rica
- Many locations, Multiple Locations, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Wu L, Bordon AF, Charles M, Rodriguez FJ, Lee J, Machewitz T, Mueller M, Del Carmen Gay G, Fromow-Guerra J; AQUILA investigators. Intravitreal aflibercept for the treatment of patients with neovascular age-related macular degeneration in routine clinical practice in Latin America: the AQUILA study. Int J Retina Vitreous. 2022 Oct 18;8(1):76. doi: 10.1186/s40942-022-00425-w. PMID 36258240
- [Derived] Rodriguez FJ, Wu L, Bordon AF, Charles M, Lee J, Machewitz T, Mueller M, Gay GDC, Fromow-Guerra J; AQUILA Investigators. Intravitreal aflibercept for the treatment of patients with diabetic macular edema in routine clinical practice in Latin America: the AQUILA study. Int J Retina Vitreous. 2022 Aug 2;8(1):52. doi: 10.1186/s40942-022-00396-y. PMID 35918743